CLINICAL TRIAL: NCT01397981
Title: Evaluation of Haptic Technologies for Movement Retraining
Brief Title: Gait Retraining to Reduce Knee Osteoarthritis Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Pete Bradley Shull, Dr., Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-07142011-8086
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Walking modification (Experimental): Changing kinematics for walking
  Interventions: Behavioral: Gait retraining

INTERVENTIONS:
Behavioral: Gait retraining — Changing the kinematics of walking

SUMMARY:
The purpose of this study is to determine how well people can be trained to produce new and different movements through the use of haptic feedback. One particular application is retraining individuals to walk differently in order to reduce knee joint loads to prevent or treat knee osteoarthritis as an alternative to surgical treatments.

DETAILED DESCRIPTION:
During the movement retraining session, you be given different combinations of haptic, visual, and auditory feedback in order to inform you on desired movement changes. This will take place at the Human Performance Laboratory at Stanford University. Motion analysis will be done while you perform movement activities (such as locomotion).

Prior to performing these movement tasks the investigators will attach reflective markers to your body using tape, pre-wrap and/or ace bandages. The investigators will record motion of your body's movements using infrared cameras which capture anatomical data from the reflective markers on your body.

The investigators will provide you with feedback to inform you of desired movement modifications. Haptic feedback devices such as vibration motors and skin stretch devices will be attached to your body via velcro straps and will be used to give "touch" feedback. There will be a computer monitor in front of you during testing to provide visual feedback. Sounds will be played using speakers near the testing area to provide auditory feedback.

The time needed for set up and performance of the above set of tests is approximately 90 minutes. You will be performing walking and other movements for only a small part of that time. The rest of the time will be spent preparing you for the experiment. After the investigators examine your movement data, if some of the data appear inaccurate or the investigators are unable to process the data, the investigators may ask you to repeat the movement analysis at a later time.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of medial compartment pain during the previous 6 weeks
* Radiographic evidence (AP X-ray) of medial compartment knee osteoarthritis (KL score of 3 or less)
* Ability to walk unaided for 25 minutes without rest
* Age > 18

Exclusion Criteria:

* BMI > 30
* Previous injury or surgery on foot, ankle, knee, hip, or back inhibiting ability to adopt different walking gait
* Use of shoe insert or hinged knee brace
* Corticosteroid injection within the previous 6 weeks
* Age > 80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Measure: Knee pain and function | four weeks
  Knee pain and function will be assessed through the standardized KOOS survey

SECONDARY OUTCOMES:
Learning retention, knee adduction moment | four weeks
  Learning retention of gait kinematics and knee joint loading including the knee adduction moment will be measured through motion capture and ground reaction force plates

CONTACTS AND LOCATIONS:
Overall Officials: Pete B Shull, Study Director — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Shull PB, Lurie KL, Cutkosky MR, Besier TF. Training multi-parameter gaits to reduce the knee adduction moment with data-driven models and haptic feedback. J Biomech. 2011 May 17;44(8):1605-9. doi: 10.1016/j.jbiomech.2011.03.016. Epub 2011 Apr 2. PMID 21459384
- [Background] Wheeler JW, Shull PB, Besier TF. Real-time knee adduction moment feedback for gait retraining through visual and tactile displays. J Biomech Eng. 2011 Apr;133(4):041007. doi: 10.1115/1.4003621. PMID 21428681
- [Result] Shull PB, Shultz R, Silder A, Dragoo JL, Besier TF, Cutkosky MR, Delp SL. Toe-in gait reduces the first peak knee adduction moment in patients with medial compartment knee osteoarthritis. J Biomech. 2013 Jan 4;46(1):122-8. doi: 10.1016/j.jbiomech.2012.10.019. Epub 2012 Nov 10. PMID 23146322